CLINICAL TRIAL: NCT06923306
Title: Virtual Reality Exposure for Vaginismus: A Replicated Single-Case Design
Acronym: VIVID 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lori Brotto, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H24-01258
Record Dates: First submitted 2025-03-25; First posted 2025-04-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-03

CONDITIONS: Vaginismus
Keywords: virtual reality; digital health; sexual health
MeSH Terms: conditions — Vaginismus | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: This study uses a multiple baseline single case design (SCD) in which the investigators will compare no treatment with VRE using a non-concurrent randomized single case A-B phase design, with 4 cohorts of 5 participants (n=20). To establish an experimental effect in SCD, ongoing assessment of outcomes throughout each phase is a necessary condition, with best-practice guidelines mandating at least 3 observations per outcome variable per phase.
  Here, for each participant, primary and secondary outcomes will be assessed repeatedly during baseline (i.e., Baseline and Psychoeducation - Phase A, lasting 1.5 - 3.5 weeks, and during Virtual Reality Exposure therapy - Phase B), lasting 3 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality exposure plus psychoeducation (Experimental): The investigators designed the VRE protocol based on interviews from our proof-of-concept study. Participants will take part in 3 x 2-hour sessions over a 3-week period. Treatment will adhere to three key principles: (i) Exposure will be prolonged, such that participants will use a VR headset to view a sexual scene multiple times; (ii) Treatment will proceed gradually, with the sexual activities depicted moving from non-penetrative (low fear) to penetrative (high fear); and (iii) Exposures will be repeated, with participants re-watching the videos until their fear response has habituated (i.e., level of distress = 10-20/100).
  Prior to their first VRE session, participants will be given access to a website with descriptions and images of a variety of VR sexual videos, which will allow them to select an exposure film based on comfort with/attraction to the virtual actor.
  Interventions: Behavioral: Virtual reality exposure

INTERVENTIONS:
Behavioral: Virtual reality exposure — This is a single case design and there is only one intervention. In the no-treatment arm, participants will only have assessment but no virtual reality exposure therapy.

SUMMARY:
Vaginismus is a sexual dysfunction characterized by involuntary tightening of the pelvic floor muscles, preventing vaginal intercourse. It is defined by an intense fear of vaginal penetration, leading to persistent difficulties with vaginal intercourse and gynaecological exams. Psychological factors play a significant role in vaginismus. If the pelvic floor muscle tightening represents a defensive reflex, then treatment using a gradual exposure to feared stimuli using virtual reality may lead to an extinction of the phobic response, and to amelioration of vaginismus. If effective, the use of virtual reality technology can directly improve clinical care offered to those suffering from vaginismus.

DETAILED DESCRIPTION:
Purpose/Aims:

VR is a new, powerful technology that, if effective, can directly improve clinical care offered to those suffering from vaginismus across Canada. This study will advance health-related knowledge by providing new data on the efficacy of VRE for vaginismus and health outcomes by having the potential to increase access to effective treatment for women living in rural and remote areas as well as those who experience other barriers in accessing care-including extreme fear or anxiety. Thus, this research program has a high likelihood of filling a major gap in healthcare for women and others with a vagina and, if effective, our treatment paradigm has significant potential for scale-up.

Hypothesis:

The investigators will use the Marascuilo-Busk randomization test to test our hypothesis that the onset of VRE leads to an increase in vaginal insertion ease, a decrease in insertion pain, and an increase in the frequency of sexual activity that includes penetration.

Justification:

Lack of Effective Treatments: Available psychological treatments for vaginismus involve self-insertion of vaginal accommodators (which resemble dildos) at home by progressively inserting larger sizes as the individual practices relaxation exercises that address both the psychological fear and the involuntary pelvic floor muscle tension. However, individuals with vaginismus experience significant and longstanding avoidance and struggle to complete accommodator exercises on their own at home, even if they believe the treatment will be effective. This avoidance significantly limits treatment effectiveness. For example, the largest RCT (n=117) evaluating the efficacy of cognitive behavioural therapy for vaginismus, which included gradual self-insertion of accommodators into the vagina, yielded a small treatment effect: only 14% of women who attended ten 2-hour group therapy sessions were able to have vaginal intercourse at post-treatment.

Exposure - An Essential Treatment Element: Therapist-guided exposure therapy includes a patient progressively inserting vaginal accomodators in the presence of a supportive clinician, and is highly effective in treating vaginismus, showing greater success than solo, self-guided interventions. Of 77 women who attended two therapist-guided sessions over one week, 89% reported vaginal intercourse 6-weeks post-treatment. Despite this effective treatment approach, in North America therapist-aided exposure practices are not permitted due to institutional restrictions, licensing regulations, and/or patient discomfort. As such, the development of alternative exposure-based treatments is needed. The investigators propose an innovative application of VR, as an alternative to exposure, to address this significant health gap.

VR Exposure - An Opportunity: VRE immerses individuals in 3D simulations of feared situations and is as effective as real-life exposure for specific phobias. VRE for vaginismus, which involves gradual exposure to feared (virtual) sexual encounters, may diminish phobic responses towards vaginal penetration. Given that women with vaginismus cope via longstanding avoidance, and often do not perform at-home exposure exercises included in frontline recommended treatments, the "immersive" nature of VRE can directly target this avoidance.

Proof of Concept: In 2022, the investigators conducted a proof-of-concept study in which they assessed the acceptability and feasibility of VRE for vaginismus. Our results indicated that patients with vaginismus experienced greater distress when viewing VR erotica and were more likely to use anxiety management strategies than controls. Despite this, 95% of participants with vaginismus endorsed VRE as an acceptable treatment option.

Theoretical Approach/Framework Fear in the Context of Genital Pain: Fear of pain elicits a cascade of cognitive-motivational and physio¬logical processes that interact with one another and influence pain processing via multiple pathways. Specifically, fear induces hypervigilance to (potentially) pain-inducing sexual stimuli, their appraisal as threatening, and draws attention away from sexually exciting cues. Negative appraisals of sexual stimuli paired with reduced attention to sexual cues inhibits genital arousal, which increases pelvic floor muscle tension and vaginal dryness. These physical changes cause mechanical friction, and in turn, pain. The association between pain and sexual activity leads to avoidance of sexual encounters. Therefore, tackling fear is a key piece of the genital pain puzzle.

Fear Learning as a Treatment Target: Research suggests that fear of genital pain is learned through classical conditioning when a neutral stimulus is paired with pain. For example, if an adolescent inserts a tampon for the first time and there is significant pain, they will learn to expect pain on subsequent insertions. As a result, they may avoid using tampons, which they think will prevent pain and/or reduce fear, reinforcing the avoidance behaviour. Their behavioural response maintains the tampon's threat value, as the absence of the painful outcome is attributed to the avoidance. In the case of vaginismus, fear generalization occurs, such that the adolescent's expectation of pain and consequent fear spreads to any type of stimulus that involves vulvar and/or vaginal touch, such as vaginal inter¬course and gynaecological exams, giving rise to a broader penetration-pain association that extends from tampons to all insertive objects.

Since fear acquisition and (especially) fear generalization play key roles in the development and maintenance of chronic genital pain, effective treatments require fear extinction via conditioning, commonly referred to as exposure therapy. Traditionally, this involves repeatedly exposing an individual to the fear-inducing stimulus until their fear decreases (habituates), which represents a corrective experience. However, recent work from experts in the study of anxiety disorders suggests that expectancy violation and inhibitory learning are the key mechanisms of exposure, with more robust treatment effects when there is a discrepancy between expected and actual outcomes. When exposure is successful, extinction does not erase the original penetration-pain association that was learned during acquisition, but a new inhibitory penetration-no pain association develops and inhibits the retrieval of the original acquisition memory.

The protocol proposed here will incorporate psychoeducation about these concepts before VRE treatment begins, repeated exposure to virtual sexual scenarios, and progressive insertion of vaginal accommodators for sensory-motor feedback training. Psychoeducation is an evidence-based intervention that provides information and support to individuals. It has been found to be beneficial when coupled with other treatments, and may be particularly important for e-health interventions. VRE treatment studies for anxiety disorders often include patient psychoeducation, VR technology, and use safety behaviours. Psychoeducational interventions for vaginismus have also proved beneficial for fear behaviours and overall well-being. Communication exercises, relaxation techniques, and sex education are common elements of these programs. The investigators predict that these treatment elements will promote the extinction of penetration-related fears for individuals with vaginismus.

ELIGIBILITY:
Inclusion Criteria:

The investigators will recruit individuals who have a vagina. They expect that most participants will identify as cisgender, where sex is female and gender is woman, while others may have a female sex but identify as a different gender (e.g., genderdiverse). Transwomen (i.e., birth assigned males but identify as woman) who have had gender-affirming surgery (and so have a vagina) are eligible, as are transmen (i.e., birth assigned females but identify as men) who have not had bottom surgery (so have a vagina).

Inclusion criteria: In addition to having a vagina, participants must have a diagnosis of vaginismus that requires self-reported involuntary tightness of the vaginal musculature that causes persistent interference with vaginal penetration lasting >6 months; aged >19 y, of any sexual orientation. Participants must be fluent in English (psychoeducational materials and questionnaires delivered in English), have normal or corrected-to-normal vision (to view the VR scenes during exposure), and be able to travel to Vancouver.

Exclusion Criteria:

Presence of: unprovoked vaginal pain; a vulvar skin condition (i.e., lichen sclerosus); an imperforate hymen; or epilepsy characterized by photosensitive seizures. Note: provoked vulvar pain is not an exclusion criterion because at least 40% of people with vaginismus report pain with attempted penetration.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Ease of vaginal insertion | Assessed 2x per week during no treatment (Phase A) and Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups.
  Ease of vaginal insertion will be measured using a modified version of the Tampon Test used extensively in Provoked Vestibulodynia research.It involves having the participant insert a small vaginal accommodator (approximately the size of a tampon) into their vagina, and rate the ease of insertion on an 11-point scale ranging from 0 (unable to insert - too difficult) to 10 (can insert with great ease).

SECONDARY OUTCOMES:
Insertion pain | Assessed 2x per week during no treatment (Phase A) and Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups.
  Insertion pain will be assessed using the Tampon Test at the same time they are assessing ease of vaginal insertion; participants will self-report their insertion pain on an 11-pt scale ranging from 0 (no pain) to 10 (worst possible pain).
Frequency of sexual activity that includes vaginal insertion | Assessed the day before Treatment (VRE - Phase B), final day of Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups.
  Participants will answer the following two questions the day before Treatment (VRE - Phase B), final day of Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups: 1. "In the past 3 weeks, have you engaged in any sexual activity that involved penetration?" Answer will be on a 3-point scale: 0 = I have not attempted to engage in sexual activity that included penetration; 1 = I have inserted my own finger or sex toy into my vagina; 2 = my partner has inserted a finger, sex toy, or penis into my vagina. 2. "How many times have you engaged in any sexual activity that involved penetration?"
Frequency of vaginal accommodator/dilator use | Assessed day before Treatment (VRE - Phase B), final day of Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups.
  Participants will answer the following two questions the day before Treatment (VRE - Phase B), final day of Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups: 1. "In the past 3 weeks, have you attempted to insert vaginal accommodators/dilators outside of the context of the study (i.e., not for ease of insertion or pain with insertion assessment?" Participants will be invited to select either: 0 = I have not attempted to insert a vaginal accommodator/dilator; 1 = I have attempted to insert a vaginal accommodator/dilator. 2. "How often have you attempted to insert vaginal accommodators/dilators outside of the context of the study (i.e., not for ease of insertion or pain with insertion assessment?"
Negative and catastrophic penetration-related cognitions (VPCQ) | Assessed day before Treatment (VRE - Phase B), final day of Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups.
  Negative and catastrophic penetration-related cognitions, will be assessed using the Vaginal Penetration Cognition Questionnaire (VPCQ), validated for vaginismus. Individuals will rate the applicability of 40 statements (e.g., I am afraid that my vagina is too narrow for penetration) using a 7-pt scale ranging from 1 (not at all applicable) to 7 (very strongly applicable).
Sexual distress (FSDS-R) | Assessed day before Treatment (VRE - Phase B), final day of Treatment (VRE - Phase B), and once at 3-weeks and 3-month follow-ups.
  Sexual distress will be measured by the Female Sexual Distress Scale-Revised (FSDS-R), used extensively in sexuality treatment outcome studies. Participants will rate 13 statements using a 5-pt numeric scale ranging from 0 (never) to 4 (always) to indicate how often they experience distress related to sexual problems.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brotto, PhD, RPsych, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - UBC Sexual Health Lab, Vancouver Hospital, Vancouver, British Columbia
  - Diamond Health Care Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
We will be providing all IPD that underlie results in a publication. We will provide Analytic Code only in addition to the data and data dictionaries. Other information will be presented in the publications or available upon request from the main author or PI.
Supporting Information: Analytic Code
Time Frame: The data will be made available within 3 months after publication.
Access Criteria: The data will be freely available on the OSF website so no need for requests.

REFERENCES:
- [Background] Milani S, Jabs F, Brown NB, Zdaniuk B, Kingstone A, Brotto LA. Virtual Reality Erotica: Exploring General Presence, Sexual Presence, Sexual Arousal, and Sexual Desire in Women. Arch Sex Behav. 2022 Jan;51(1):565-576. doi: 10.1007/s10508-021-02111-8. Epub 2021 Oct 25. PMID 34697691
- [Background] Wechsler TF, Kumpers F, Muhlberger A. Inferiority or Even Superiority of Virtual Reality Exposure Therapy in Phobias?-A Systematic Review and Quantitative Meta-Analysis on Randomized Controlled Trials Specifically Comparing the Efficacy of Virtual Reality Exposure to Gold Standard in vivo Exposure in Agoraphobia, Specific Phobia, and Social Phobia. Front Psychol. 2019 Sep 10;10:1758. doi: 10.3389/fpsyg.2019.01758. eCollection 2019. PMID 31551840
- [Background] Ter Kuile MM, Melles R, de Groot HE, Tuijnman-Raasveld CC, van Lankveld JJDM. Therapist-aided exposure for women with lifelong vaginismus: a randomized waiting-list control trial of efficacy. J Consult Clin Psychol. 2013 Dec;81(6):1127-1136. doi: 10.1037/a0034292. Epub 2013 Sep 23. PMID 24060195